



Acute Effects of Endurance Exercise with Moderate and High Intensity on Breast Milk Composition Among Women with Overweight/Obesity

Acronym: YT

NCT number: NCT05745922

Document date: 02. January 2024

Document type: Informed consent partner (Translated from Norwegian)







## REQUEST FOR CONSENT TO THE COLLECTION OF INFORMATION ABOUT YOUR CHILD IN THE RESEARCH PROJECT

# Acute effects of moderate and high intensity endurance training on breast milk composition

Since your partner is participating in a research project where we are investigating the effect of two different training sessions on breast milk composition, you are asked to consent to the collection of information about your baby. The study is being conducted at NTNU in collaboration with St. Olavs Hospital.

#### WHAT DOES THE PROJECT MEAN FOR YOU?

The project involves recording information about your baby (birth weight, length, head circumference, gender). At the start of the study, we will weigh the baby, measure how long it is and examine the baby's body composition using bioimpedance.

In the project, we will collect and record information about your child. This includes: the baby's gender, information about weight, length and head circumference at birth, and the baby's weight, length and body composition at the start of the study.

#### POSSIBLE ADVANTAGES AND DISADVANTAGES

There are no specific advantages or disadvantages for you by consenting to the collection.

#### VOLUNTARY PARTICIPATION AND POSSIBILITY TO WITHDRAW YOUR CONSENT

Giving consent is voluntary. If you agree to us collecting information from your child, sign the consent form on the last page. You can withdraw your consent at any time without giving any reason. There will be no negative consequences for the child's possible treatment if you do not want to give consent or if you later wish to withdraw it. If you withdraw your consent, no further research will be conducted on the child's health information. You can request access to the information stored about the child, and the information will then be provided within 30 days. You can also request that the child's health information in the project be deleted. The right to request deletion or provision does not apply if the information has been anonymized or published. This right may also be limited if the information has been included in analyses performed.

If you later wish to withdraw your consent or have questions about the project, you can contact project manager Trine Moholdt by telephone at 97098594 or trine.moholdt@ntnu.no.

#### WHAT HAPPENS TO YOUR CHILD'S INFORMATION?

The information registered about your child will only be used as described above in the purpose of the project. You have the right to access the information registered about your child and the right to have any errors in the registered information corrected. You also have the right to access the secure measures when processing the information.





Version 3.0, 02. januar 2024

All information will be processed without name and personal identification number or other directly identifiable information. A code links you to information about your child through a list of names. Only project manager Trine Moholdt, doctoral fellows Mäeliss Limoine and Emily Rose Ashby, medical student Rebecca Holm, and project employee Guro Rosvold have access to this list.

#### INFORMATION SHARING AND TRANSFER ABROAD

By participating in the project, you also agree that all the information we collect in the project may be delivered abroad as part of research collaboration and publication. The project manager will ensure that your information is handled in a secure manner. NTNU is responsible for ensuring that the transfer of information is in accordance with Norwegian law and the EU's data protection legislation (GDPR). The code that links the child to personally identifiable information will not be disclosed abroad. As part of making research more open, we also want to share the analysis results openly with other researchers. This sharing will be de-identified. You can choose whether you want to consent to your child's data being included in such open sharing on the consent form on the last page.

#### **INSURANCE**

Participants are covered by the Patient Injuries Act.

#### **APPROVALS**

The Regional Committee for Medical and Health Research Ethics has assessed the project and has given prior approval. Case no. at REK is 562012

According to the new Personal Data Act, the controller NTNU and project manager Trine Moholt has an independent responsibility to ensure that the processing of information about your child has a legal basis. This project has a legal basis in the EU General Data Protection Regulation, Article 6, No. 1a and Article 9, No. 2a and your consent.

You have the right to complain about the processing of information about your child to the Norwegian Data Protection.

#### CONTACT INFORMATION

If you have any questions about the project, please contact Trine Moholdt, 97098594, trine.moholdt@ntnu.no.

You can contact the institution's data protection officer if you have any questions about the processing of your child's personal data in the project. NTNU's data protection officer is Thomas Helgesen, 93079038, personvernombud@ntnu.no.





### I CONSENT TO MY CHILD'S PERSONAL INFORMATION BEING USED AS DESCRIBED

| Please cross one of the two boxes below: | |
|---|---|
| I also agree that my child's data is included in the | open sharing of analysis results. |
| I do NOT consent to my child's data being include | d in the open sharing of analysis results. |
| Place and date | Guardian's signature |
| | Guardian's name in capital letters |